CLINICAL TRIAL: NCT04285307
Title: The Effect of Sleep Extension in Teenage Girls at a College Preparatory High School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Divine Savior Holy Angels High School (Unknown); Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Louella Amos, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1176849
Record Dates: First submitted 2020-01-01; First posted 2020-02-26 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2021-12

CONDITIONS: Sleep Hygiene; Sleep
Keywords: Actigraphy; Sleep Extension
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): Study group
  Interventions: Behavioral: Sleep Hygiene tips

INTERVENTIONS:
Behavioral: Sleep Hygiene tips — Students receive a packet of information on how to improve their sleep habits and hygiene.

SUMMARY:
If teenagers attain the recommended amount of sleep (9-9.5 hours per night), they will feel less stress and have better athletic and academic performance.

The investigators will track students sleep patterns before and after a sleep intervention where they are given a packet of sleep tips and encouraged to improve their sleep hygiene.

Outcomes include stress levels, academic/athletic performance, and sleep cycle data from the sleep tracking watch.

DETAILED DESCRIPTION:
A. PURPOSE OF THE STUDY

To determine the effect of sleep extension on stress levels, cognitive function, and fitness in teenage girls.

B. HYPOTHESIS / SPECIFIC AIMS

If teenagers attain the recommended amount of sleep (9-9.5 hours per night), they will feel less stress and have better athletic and academic performance.

Primary Objective:

• The investigators will evaluate stress with a validated questionnaire before and after sleep extension (increased total sleep time per night).

Secondary Objectives:

* The investigators will evaluate physical fitness and endurance with standardized testing before and after sleep extension.
* The investigators will measure several sleep variables (total sleep time, sleep efficiency, sleep onset latency, sleep-wake cycle pattern, sleepiness) before and after sleep extension.
* The investigators will evaluate the association between academic performance (Grade Point Average (GPA) and average total sleep time per night.

Intervention:

Sleep extension: Increasing nightly total sleep time (goal of 9-9.5 hours per night) by improving sleep hygiene, daily exercise, etc.

In a prospective cohort study, up to 40 otherwise healthy teenage girls age 14-18 years at DSHA High School will be approached for consent to participate in the study. Upon consent they will complete the Insomnia Severity Index (ISI), Epworth Sleepiness Scale for Children and Adolescents (ESS-ChAD) and Perceived Stress Scale (PSS) questionnaires and will be issued an actigraphy watch to monitor their sleep-wake cycles daily at home for 2 weeks. They will also keep a sleep diary during the study period.

After the 2 weeks of actigraphy, subjects will have the data from the actigraphy watch downloaded and submit their sleep diary. They will be given sleep hygiene recommendations to try to attain 9-9.5 hours of sleep per night (sleep extension), if not already sleeping this amount. They will then be given a different actigraphy watch to wear and another sleep diary to log their total sleep time for 4 more weeks.

After the 4 weeks, the actigraphy watch will be returned, the actigraphy data will be downloaded and the sleep diary data will be collected. Subjects will complete the ESS-ChAD and PSS upon conclusion of the study. Subjects will be offered a report of their sleep and activity data after completing the sleep extension period. If there is a gap of more than 4 weeks between actigraphy use and the second fitness test, the investigators will ask participants to complete another 1-week sleep diary prior to testing. All study activities except downloading the actigraphy watch data will occur at Divine Savior Holy Angels High School (DSHA).

ELIGIBILITY:
Inclusion Criteria:

1. Female students age 14-18 yrs (DSHA students ranging from Freshman to Senior year)

Exclusion Criteria:

1. Subjects and/or parent/guardian unable to read, understand or speak English
2. Subjects unable to undergo fitness testing
3. Subjects who are pregnant or become pregnant during the course of the study

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Stress Levels | Week 0 (before actigraphy) and Week 6 (after both actigraphy watch courses)
  Perceived Stress Scale (PSS); 10 questions, scores between 0-4; higher score shows higher stress levels

SECONDARY OUTCOMES:
Change in Physical Fitness | 6 months (end of August to end of February)
  Standardized PACER (Progressive Aerobic Cardiovascular Endurance Run) testing; administered in the Fall and Spring of each school year; a series of timed runs that get progressively faster; Out of 25 laps, higher score is better with more laps completed
Sleepiness | 6 weeks, 2 before intervention and 4 after
  Difference in sleepiness before and after sleep extension intervention. Measured with the Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD); scale of 0 to 3; higher score means more likely to fall asleep in a given situation
Total Sleep Time | 6 weeks, 2 before intervention and 4 after
  Difference in total sleep time before and after sleep extension intervention
Sleep Latency | 6 weeks, 2 before intervention and 4 after
  Difference in sleep latency before and after sleep extension intervention
Academic performance | First semester 4 months (August 19th, 2019 - December 20th, 2019)
  Grade point average (GPA); 0.0-4.0 scale, higher is better

CONTACTS AND LOCATIONS:
Locations (1):
- Divine Savior Holy Angels High School, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carskadon MA, Harvey K, Duke P, Anders TF, Litt IF, Dement WC. Pubertal changes in daytime sleepiness. 1980. Sleep. 2002 Sep 15;25(6):453-60. No abstract available. PMID 12224838
- [Background] Wolfson AR, Carskadon MA. Sleep schedules and daytime functioning in adolescents. Child Dev. 1998 Aug;69(4):875-87. PMID 9768476
- [Background] Lee YJ, Park J, Kim S, Cho SJ, Kim SJ. Academic performance among adolescents with behaviorally induced insufficient sleep syndrome. J Clin Sleep Med. 2015 Jan 15;11(1):61-8. doi: 10.5664/jcsm.4368. PMID 25515277
- [Background] Mah CD, Mah KE, Kezirian EJ, Dement WC. The effects of sleep extension on the athletic performance of collegiate basketball players. Sleep. 2011 Jul 1;34(7):943-50. doi: 10.5665/SLEEP.1132. PMID 21731144
- [Background] Schwartz J, Simon RD Jr. Sleep extension improves serving accuracy: A study with college varsity tennis players. Physiol Behav. 2015 Nov 1;151:541-4. doi: 10.1016/j.physbeh.2015.08.035. Epub 2015 Sep 1. PMID 26325012
- [Background] Adolescent Sleep Working Group; Committee on Adolescence; Council on School Health. School start times for adolescents. Pediatrics. 2014 Sep;134(3):642-9. doi: 10.1542/peds.2014-1697. PMID 25156998
- [Background] National Sleep Foundation. Eight major obstacles to delaying school start times. http://sleepfoundation.org/sleep-news/eight-major-obstacles-delaying-school-start-times.
- [Background] Janssen KC, Phillipson S, O'Connor J, Johns MW. Validation of the Epworth Sleepiness Scale for Children and Adolescents using Rasch analysis. Sleep Med. 2017 May;33:30-35. doi: 10.1016/j.sleep.2017.01.014. Epub 2017 Feb 12. PMID 28449902
- [Background] Kanady JC, Drummond SP, Mednick SC. Actigraphic assessment of a polysomnographic-recorded nap: a validation study. J Sleep Res. 2011 Mar;20(1 Pt 2):214-22. doi: 10.1111/j.1365-2869.2010.00858.x. PMID 20626612
- [Background] Natale V, Plazzi G, Martoni M. Actigraphy in the assessment of insomnia: a quantitative approach. Sleep. 2009 Jun;32(6):767-71. doi: 10.1093/sleep/32.6.767. PMID 19544753